CLINICAL TRIAL: NCT04076566
Title: Prospective Study in the Use of the Alfapump® in the Treatment of Malignant Ascites
Brief Title: Malignant Ascites Alfapump® Study
Acronym: ProMAS
Status: Withdrawn | Type: Observational
Why Stopped: Update to clinical strategy - COVID impact
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-AAR-013
Record Dates: First submitted 2019-08-02; First posted 2019-09-03 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2019-08

CONDITIONS: Malignant Ascites
Keywords: OVARIAN; COLORECTAL; PARACENTESIS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: alfapump system — active implantable device for treatment of malignant ascites

SUMMARY:
ProMAS is a prospective post-marketing, single-arm study to assess performance and safety of the Alfapump® system in the treatment of patients with malignant ascites. The study aims to enroll 40 patients in up to 8 sites in Europe.

DETAILED DESCRIPTION:
The Prospective Malignant Ascites Alfapump® study is a single-arm, prospective study to evaluate the performance and safety of the Alfapump® system in the treatment of patients with malignant ascites. The Alfapump® system is a fully implantable programmable pump, able to move ascitic fluid from the peritoneal cavity to the bladder via 2 catheters. The Alfapump® has obtained CE (Conformité Européenne) mark approval for the indication of malignant ascites. The primary objective of the study is to assess the performance of the system to remove ascites. Secondary objectives are to evaluate the safety and tolerability of the Alfapump® in the treatment of malignant ascites for a total follow-up period of 9 months, and to evaluate quality of life (QoL) by reduction or elimination of paracentesis requirement. Furthermore the study includes an exploratory scientific objective as to feasibility to obtain 'liquid biopsy' samples suitable for analysis in a non-invasive way after Alfapump® implantation. 40 patients with malignant ascites will be enrolled in up to 8 sites in Europe (Belgium, United Kingdom, Switzerland). Specific sub-analysis of data from patients with gynecological (ovarian) cancer is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age;
2. Subject has provided written informed consent; 3.Subject has recurrent malignant ascites defined as ≥2 therapeutic paracenteses in the month prior to enrolment; 4.Subject has sufficient baseline data documented for at least 4 paracentesis events in the last 3 months pre-implant, including date and volume; 5.Subject has ascites following neoplastic disease, as assessed by physician. In subjects with primary malignancy of the liver it should be confirmed that the ascites is due to malignancy and not due to underlying pre-existing cirrhosis.

6.Subject has a life expectancy of ≥3 months as assessed by the treating physician, and is receiving or intended to receive anticancer therapy.

7.Subject has the ability to comply with study procedures, including all follow-up visits at implanting centre when required, and ability to perform subject-required system tasks (charging). A subject with a caregiver who can comply with the study procedures and to perform the tasks required for appropriate pump function is allowed as well.

Exclusion Criteria:

1. Subject has evidence of multiple ascites loculation
2. Ascites analysis with neutrophil count >250/µl within 24-hours prior to implant.
3. Subject has acute Urinary Tract Infection (UTI) within 24-hours of implantation assessed by urinalysis.
4. Subject has skin infection of the abdominal wall at the area of implantation.
5. Subject has a serum creatinine > 1.5 mg/dL Subject has
6. Subject has obstructive uropathy (bladder residual volume >100 mL, determined by catheterization or abdominal ultrasound) in case of Lower Urinary Tract Symptoms (LUTS) .
7. Existing bladder anomaly denying proper catheterization of the bladder.
8. Subject has active bleeding or thrombocytopenia < 45,000 X106/L.
9. Subject on long-term prophylactic anticoagulation
10. Subject is pregnant or a female of childbearing potential.
11. Patient has recurrent requirement for MRI
12. Subject is currently participating in an oncology trial which might be negatively affected by the alfapump as assessed by the treating physician

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Investigators will be asked to enrol subjects meeting the inclusion and exclusion criteria .This study population is highly palliating with overall limited prognosis and significant comorbidities and possibly reduced performance status. Subjects must be under the care of an oncologist specialised in their disease. In the case of hepatic involvement, a hepatologist, and in the case of ovarian or breast cancer a gynaecologic oncologist accustomed to managing subjects with advanced malignancy. Subjects will be enrolled into the trial from the clinical practices of the investigators. Suitable subjects will undergo screening, including detailed medical history, paracentesis history and blood tests, to ensure compliance with study inclusion / exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-31 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Monthly therapeutic paracentesis frequency up to 3 months | 3 months post-implantation
  Monthly therapeutic paracentesis frequency up to 3 months compared to the baseline therapeutic paracentesis frequency.
  The monthly therapeutic paracentesis frequency up to 3 months is defined as the average rate of therapeutic paracenteses during month 1, 2 and 3 post-implantation.
  Baseline therapeutic paracentesis frequency is defined as the average rate of therapeutic paracentesis in the 3 months prior to pump implantation.

SECONDARY OUTCOMES:
Monthly therapeutic paracentesis frequency up to 6 months | 6 months post-implantation
  Monthly therapeutic paracentesis frequency up to 6 months compared to the baseline therapeutic paracentesis frequency.
  The monthly therapeutic paracentesis frequency at 6 months is defined as the average rate of therapeutic paracenteses during months 1 to 6 Baseline therapeutic paracentesis frequency is defined as the average rate of therapeutic paracentesis in the 3 months prior to pump implantation.
Safety outcome: free survival | Time (days) to first paracentesis after implantation through 270 days post implantation
  Therapeutic paracentesis free survival after Alfapump® implantation
Efficacy outcome- Assessment of changes in Quality of Life | at 1-month, 3-month, 6-month and 9-month follow-up compared to baseline
  Changes in Quality of life after Alfapump® implantation, measured with validated EORTC cancer related Quality of life Questionnaire-CR29 (ColoRectal 29 questions) in subjects with colorectal malignancy.
Efficacy outcome- Assessment of changes in Quality of Life | at 1-month, 3-month, 6-month and 9-month follow-up compared to baseline
  Changes in Quality of life after Alfapump® implantation assessed with validated FACIT-AI 5Ascites Index) ascites related quality of life questionnaire in all subjects enrolled in the study.
Efficacy outcome- Assessment of changes in Quality of Life | at 1-month, 3-month, 6-month and 9-month follow-up compared to baseline
  Changes in Quality of life after Alfapump® implantation, measured with validated EORTC-cancer related Quality of life questionnaire-OV28 (OVarian 28 questions), in subjects with a gynaecological malignancy.
Nutritional status outcome | at 1-month, 3-month, 6-month and 9-month follow-up compared to baseline
  Change in nutritional status assessed by Psoas muscle measurement
Nutritional status outcome | at 1-month, 3-month, 6-month and 9-month follow-up compared to baseline
  Change in nutritional status assessed by changes in serum Zinc
Nutritional status outcome | at 1-month, 3-month, 6-month and 9-month follow-up compared to baseline
  Change in nutritional status assessed by changes in serum pre-albumin
Nutritional status outcome | at 1-month, 3-month, 6-month and 9-month follow-up compared to baseline
  Change in nutritional status assessed by changes in serum phosphate
Nutritional status outcome | at 1-month, 3-month, 6-month and 9-month follow-up compared to baseline
  Change in nutritional status assessed by changes in serum potassium
Nutritional status outcome | at 1-month, 3-month, 6-month and 9-month follow-up compared to baseline
  Change in nutritional status assessed by changes in serum albumin
Pump performance | at 1-month, 3-month, 6-month and 9-month follow-up
  Total Monthly volume of ascitic fluid removed (sum of volumes removed during each month via either Alfapump® and via therapeutic paracentesis)
Pump performance outcome - pump survival | Time (days) from implantation until explantation due to technical causes through study completion up to 270 days post-pump implantation
  Pump survival through study completion, up to 270 days post-pump implantation
Pump performance outcome - pump survival | Time (days) from implantation until first exchange due to technical causes through study completion up to 270 days post-pump implantation
  Pump survival through study completion, up to 270 days post-implantation
Pump performance outcome | through study completion up to 270 days post-pump implantation
  Frequency of hospitalisations following Alfapump® implantation through study completion up to 270 days post-pump implantation
Pump performance outcome | throug study completion up to to 270 days post-pump implantation
  Duration of hospitalisations following Alfapump® implantation through study completion up to 270 days post-pump implantation
Safety outcome - subject survival | Time (days) until exitus through study completion up to 270 days post-pump implantation
  Subject overall survival after Alfapump® implantation through study completion up to 270 days post-pump implantation
Safety outcome- Bladder metastasis: Freedom from metastatic bladder wall infiltration | at 6-month follow-up
  Freedom from metastatic bladder wall infiltration as assessed by cystoscopy
Safety outcome- Worsening of renal function | at 3-month, 6-month and 9-month follow-up compared to baseline
  Incidence of subjects suffering Renal function deterioration, defined as a rise in serum creatinine of ≥50% or ≥0.3mg/dl .
Safety outcome- Incidence of device related infection | at 3-month, 6-month and 9-month follow-up
  Incidence of Device-related infections following pump-implantation
Safety outcome- Incidence of Procedure related events | At 1 month follow-up.
  Incidence of Procedure related adverse events
Safety outcome- Incidence of Device related events | at 3-month, 6-month and 9-month follow-up
  Incidence of any Device-related adverse events
Device failure | Through study completion up to 270 days post-pump implantation
  Incidence of device failure resulting in re-intervention (Revision, exchange or explantation) through study completion up to 270 days post-pump implantation

OTHER OUTCOMES:
Exploratory outcome- liquid biopsies | 2-days, 7-days, 3-months, 6-months and 9-months post implant
  Incidence of successful acquisition of ascitic fluid samples appropriate for oncological analysis via Alfapump® function
Exploratory outcome - anticancer treatment | Time (days) to event through study completion up to 270 days post-pump implantation
  Incidence of Initiation of new / change to existing anticancer treatment through study completion up to 270 days post-pump implantation

CONTACTS AND LOCATIONS:
Overall Officials: Christina Fotopoulou, Prof, MD, Principal Investigator — Imperial Hospital, London, UK
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers

REFERENCES:
- [Background] European Association for the Study of the Liver. EASL clinical practice guidelines on the management of ascites, spontaneous bacterial peritonitis, and hepatorenal syndrome in cirrhosis. J Hepatol. 2010 Sep;53(3):397-417. doi: 10.1016/j.jhep.2010.05.004. Epub 2010 Jun 1. No abstract available. PMID 20633946
- [Background] Pache I, Bilodeau M. Severe haemorrhage following abdominal paracentesis for ascites in patients with liver disease. Aliment Pharmacol Ther. 2005 Mar 1;21(5):525-9. doi: 10.1111/j.1365-2036.2005.02387.x. PMID 15740535
- [Background] Lin CH, Shih FY, Ma MH, Chiang WC, Yang CW, Ko PC. Should bleeding tendency deter abdominal paracentesis? Dig Liver Dis. 2005 Dec;37(12):946-51. doi: 10.1016/j.dld.2005.07.009. Epub 2005 Sep 26. PMID 16185942
- [Background] Gines P, Tito L, Arroyo V, Planas R, Panes J, Viver J, Torres M, Humbert P, Rimola A, Llach J, et al. Randomized comparative study of therapeutic paracentesis with and without intravenous albumin in cirrhosis. Gastroenterology. 1988 Jun;94(6):1493-502. doi: 10.1016/0016-5085(88)90691-9. PMID 3360270
- [Background] Sola R, Vila MC, Andreu M, Oliver MI, Coll S, Gana J, Ledesma S, Gines P, Jimenez W, Arroyo V. Total paracentesis with dextran 40 vs diuretics in the treatment of ascites in cirrhosis: a randomized controlled study. J Hepatol. 1994 Feb;20(2):282-8. doi: 10.1016/s0168-8278(05)80070-4. PMID 7516361
- [Background] Gines A, Fernandez-Esparrach G, Monescillo A, Vila C, Domenech E, Abecasis R, Angeli P, Ruiz-Del-Arbol L, Planas R, Sola R, Gines P, Terg R, Inglada L, Vaque P, Salerno F, Vargas V, Clemente G, Quer JC, Jimenez W, Arroyo V, Rodes J. Randomized trial comparing albumin, dextran 70, and polygeline in cirrhotic patients with ascites treated by paracentesis. Gastroenterology. 1996 Oct;111(4):1002-10. doi: 10.1016/s0016-5085(96)70068-9. PMID 8831595
- [Background] MEDDEV 2.12-1, rev 7, Guidelines on a medical device vigilance system.
- [Background] Bureau C, Adebayo D, de Rieu MC, Elkrief L, Valla D, Peck-Radosavljevic M, McCune A, Abbadi R, Vargas V, Simon-Talero M, Cordoba J, Angeli P, Rosi S, MacDonald S, Malago M, Stepanova M, Younossi ZM, Trepte C, Watson R, Borisenko O, Sun S, Inhaber N, Jalan R. Corrigendum to "Alfapump(R) system vs. large volume paracentesis for refractory ascites: A multicenter randomized controlled study" [J Hepatol 67 (2017) 940-949]. J Hepatol. 2018 Mar;68(3):630. doi: 10.1016/j.jhep.2017.12.017. Epub 2018 Feb 1. No abstract available. PMID 29395458
- [Background] Stirnimann G, Berg T, Spahr L, Zeuzem S, McPherson S, Lammert F, Storni F, Banz V, Babatz J, Vargas V, Geier A, Stallmach A, Engelmann C, Trepte C, Capel J, De Gottardi A. Treatment of refractory ascites with an automated low-flow ascites pump in patients with cirrhosis. Aliment Pharmacol Ther. 2017 Nov;46(10):981-991. doi: 10.1111/apt.14331. Epub 2017 Sep 21. PMID 28940225
- [Background] Lai JC, Covinsky KE, Dodge JL, Boscardin WJ, Segev DL, Roberts JP, Feng S. Development of a novel frailty index to predict mortality in patients with end-stage liver disease. Hepatology. 2017 Aug;66(2):564-574. doi: 10.1002/hep.29219. Epub 2017 Jun 28. PMID 28422306
- [Background] Chang L, Ni J, Zhu Y, Pang B, Graham P, Zhang H, Li Y. Liquid biopsy in ovarian cancer: recent advances in circulating extracellular vesicle detection for early diagnosis and monitoring progression. Theranostics. 2019 May 31;9(14):4130-4140. doi: 10.7150/thno.34692. eCollection 2019. PMID 31281536
- [Background] Palmirotta R, Lovero D, Cafforio P, Felici C, Mannavola F, Pelle E, Quaresmini D, Tucci M, Silvestris F. Liquid biopsy of cancer: a multimodal diagnostic tool in clinical oncology. Ther Adv Med Oncol. 2018 Aug 29;10:1758835918794630. doi: 10.1177/1758835918794630. eCollection 2018. PMID 30181785
- [Background] Giannopoulou L, Kasimir-Bauer S, Lianidou ES. Liquid biopsy in ovarian cancer: recent advances on circulating tumor cells and circulating tumor DNA. Clin Chem Lab Med. 2018 Jan 26;56(2):186-197. doi: 10.1515/cclm-2017-0019. PMID 28753534